CLINICAL TRIAL: NCT04249245
Title: Role of Nasal Dysbiosis in Parkinson Disease
Acronym: SMELLPARK
Status: Completed | Type: Observational
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-030
Record Dates: First submitted 2020-01-20; First posted 2020-01-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Parkinson Disease
Keywords: Olfaction; Microbiota; Dysbiosis; Metagenomic analysis
MeSH Terms: conditions — Parkinson Disease; Anosmia; Dysbiosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Nasal bacterial swab sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson Patients: These patients are Hospitalized or consult in the participating hospitals of the Pointe à Pitre (Guadeloupe), or at the Pitié-Salpêtrière hospital (Paris).
  They were diagnosed Idiopathic PD (Parkinson Disease). The diagnosis is made according to the MDS criteria described in Postuma and al. 2015.
  Interventions: Other: Nasal Swab
- Control Subjects: They are Spouse of Parkinson Patients group , with an age difference <5 years compared to the patient concerned.
  If the Spouse can't be included, a corresponding control subject could be recruited in the consultation with an age difference <5 years compared to the patient concerned, in respecting the final gender ratio of the PD group.
  Interventions: Other: Nasal Swab

INTERVENTIONS:
Other: Nasal Swab — All

SUMMARY:
Olfactory dysfunction is frequent in Parkinson Disease (PD) and may be present years before the motor symptoms appear. The early olfactory dysfunction could result from environmental factors acting through the nasal cavity such as microbial communities. In across-sectional bicentric study, groups of 160 PD patients and 160 controls will be compared for nasal microbiota composition according to their geographical origin. We will search an association between microbiota and the presence of an olfactory deficit, cognitive deficit and thymic disorder.

DETAILED DESCRIPTION:
Olfactory dysfunction is frequent in Parkinson Disease (PD) and may be present years before the motor symptoms appear. The early olfactory dysfunction could result from environmental factors acting through the nasal cavity such as microbial communities. Local inflammation induced by a nasal bacterial dysbiosis (microbiota imbalance) could lead to early neuronal dysfunctions in the olfactory system propagating in all the brain, thus inducing motor, cognitive and emotional manifestations in PD, in keeping with the Braak's stage hypothesis. We propose a translational project aiming at investigating the potential influence of nasal dysbiosis in PD pathogenesis. First, we will analyze both olfaction and nasal microbiota in a large series of PD patients and test the link between olfactory deficits and nasal dysbiosis. Then, we will take advantage of studying two populations of subjects with a very different environmental exposure (in mainland France and French West Indies) to isolate the abnormalities of the nasal microbiota that could be specific for PD. The study will be performed in 160 patients and 160 healthy volunteers. Patients will be enrolled in two investigators sites of which different environmental exposure: 1) Guadeloupe Hospital, French West Indies and 2) Pitie-Salpetriere Hospital, Paris, France. The patient selection will be conducted in consultation with the physician and it will be proposed to the spouse to participate as controls. When the spouse cannot be included, a corresponding witness will be recruited.The study subjects will be enrolled after collecting their informed consent.

As soon as the study subjects are included, the following measurements will be done at once at the inclusion:

* Neurological assessment: Idiopathic PD. Severity of the disease will be evaluated using the Hoehn and Yahr staging. Non-motor manifestations of the disease will be assessed using the Non-Motor Symptoms Scale (NMSS). Severity of REM behavior disorder will be evaluated using the Innsbruck REM sleep behaviour disorder inventory .
* Olfactory function: Olfactory performance will be measured using (a) the Sniffin' Stick test battery (Burghardt, Wedel, Germany) following a standardized procedure and (b) a discrimination test of odorant mixtures developed by the Research Unit.
* Global cognitive performance and executive functions: The Montreal Cognitive Assessment (MoCA) will be used to assess global cognitive performance. Frontal Assessment Battery (FAB) will be used to detect executive dysfunction.
* Memory: The delayed paragraph recall index from the Wechsler Memory Scale IV-Revised will be employed as a valid, sensitive measure of verbal declarative memory and a surrogate marker of hippocampal function.
* Mood disorders: Two self-questionnaires will be used: the Snaith-Hamilton pleasure scale to assess anhedonia severity, and the Quick inventory of depressive symptomatology-self-rated for depression intensity evaluation. Two clinician rating tests for depression severity will also be used: the Hamilton Depression Rating Scale 17 and the MINI.

Sampling of human microbiota will be performed at the end. Subjects will undergo nasal brushing from anterior nares after local epinephrine application with a sterile flocked swab inserted and gently rolled around the inside of both nostrils. Swabs (one per nostril) will be placed on ice immediately after collection and then frozen at -80°C before shipment to the Research Unit (Institut Pasteur) where analyses will be carried out:

* Immunohistochemistry analysis: The levels of Neuroinflammation and aSyn proteins will be analyzed in the nasal tissue samples.
* Microbiome analysis: Microbial composition will be determined by metagenomics (microbial whole genome sequencing).

ELIGIBILITY:
Inclusion Criteria:

Patients (PD)

* Age > 18 years
* Idiopathic PD
* In Guadeloupe (N=80) : living for more than 15 years in Caribbean, including the 5 first years.
* In Paris (N=80): living for more than 15 years in mainland France, including the 5 first years.

Controls

* Age > 18 years
* Spouse of enrolled PD patient or matched controls, with age difference between spouses <5 years. When the spouse cannot be included, a matched control respecting the PD group's final sex ratio and with an age difference <5 years relative to the concerned PD case will be enrolled.

Exclusion Criteria (both PD patients and controls)

* Presence of a cold or acute pathology which could explain an original olfactory disorder other than Parkinson's disease
* Use of nasal antiseptics within the last 3 months
* Refusal of or contraindication to nasal microbiota sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parkinson patients and control subjects (spouse or matched controls)
Sampling Method: Non-Probability Sample
Enrollment: 285 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Bacterial composition of the nasal swab samples based on whole genome sequencing | 4 years
  The amplicon sequence variants (ASV) will be constructed and comparison between groups will be performed.

SECONDARY OUTCOMES:
Epidemiological characteristics of patients PD | 4 years
  Demographic variables (locations of residence and types of housing), risk factors (activities, diet, history family).
Olfactory function | 4 years
  Olfactory performance will be measured using the Sniffin' Stick test battery (Burghardt, Wedel, Germany) following a standardized procedure and a discrimination test of odorant mixtures developed by the Research Unit
Neurological assessment: Idiopathic PD - Hoehn and Yahr staging. | 4 years
  Severity of the disease will be evaluated using the Hoehn and Yahr staging.
Neurological assessment: Idiopathic PD - Non-Motor Symptoms Scale (NMSS) | 4 years
  Severity of non-motor manifestations of the disease will be assessed using the Non-Motor Symptoms Scale (NMSS).
Neurological assessment: Idiopathic PD - the Innsbruck REM sleep behaviour disorder inventory | 4 years
  Severity of REM behavior disorder will be evaluated using the Innsbruck REM sleep behaviour disorder inventory .
Global cognitive performance - MoCA | 4 years
  The Montreal Cognitive Assessment (MoCA) will be used to assess global cognitive performance.
Executive functions | 4 years
  Frontal Assessment Battery (FAB) will be used to detect executive dysfunction.
Memory Function | 4 years
  The delayed paragraph recall index from the Wechsler Memory Scale IV-Revised will be employed as a valid, sensitive measure of verbal declarative memory and a surrogate marker of hippocampal function.
Mood disorders - the Snaith-Hamilton pleasure scale | 4 years
  The Snaith-Hamilton pleasure scale (self-questionnaire) will be used to assess anhedonia severity,
Mood disorders - the Quick inventory of depressive symptomatology-self-rated | 4 years
  The Quick inventory of depressive symptomatology-self-rated will be used for depression intensity evaluation.
Mood disorders - the Hamilton Depression Rating Scale 17 | 4 years
  The Hamilton Depression Rating Scale 17, a clinician rating test, will also be used to assess depression severity.
Mood disorders - the MINI | 4 years
  The MINI, a clinician rating test, will also be used to assess depression severity.

CONTACTS AND LOCATIONS:
Locations (2):
- Pitie-Salpetriere Hospital, Paris, France
- Centre Hospitalier Universitaire, Pointe-à-Pitre, Guadeloupe